CLINICAL TRIAL: NCT06060769
Title: Study on the Quantitative Assessment of the Risk of Hepatocellular Carcinoma in Patients With Chronic Liver Disease Using Multi-parameter Magnetic Resonance Imaging
Status: Recruiting | Type: Observational
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.FSK.028
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Cirrhosis； Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — patient-derived tumor samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC group: Patients who develop HCC during follow-up
- non-HCC group: Patients who did not develop HCC during follow-up

SUMMARY:
Quantitative MRI scanning parameters such as T1 mapping, T2 mapping, T1ρ, and elastography are used, combined with clinical and laboratory indicators, to predict the risk of liver cancer in patients with cirrhosis.

DETAILED DESCRIPTION:
Retrospectively and prospectively collect T1 mapping, T2 mapping, T2* mapping, T1ρ, elastography and other multi-parameter MRI sequence images and clinical and laboratory examination data from patients with liver cirrhosis, and conduct 5-year clinical follow-up and monitoring of all enrolled patients. Whether patients develop hepatocellular carcinoma, patients are divided into liver cancer occurrence group and non-hepatocellular carcinoma group according to clinical follow-up results. Cox proportional hazard analysis is used to compare the differences in clinical characteristics, laboratory tests, imaging characteristics, quantitative MRI parameters and other variables between the two groups of patients. , and calculate the hazard ratio for each variable; assign a score to each covariate based on the proportion of the hazard ratio in the multivariable model, and develop a nomogram to predict HCC risk by the total score.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged over 18 years old; 2. Liver function Child-Pugh classification A or B; 3. Patients with chronic liver disease who meet the diagnostic criteria for high-risk groups of liver cancer in the "Guidelines for the Diagnosis and Treatment of Primary Liver Cancer (2022 Edition)"; 4. Equipped with Gd-EOB-DTPA enhanced MRI scan images, including T1 mapping, T2 mapping, T2* mapping, T1ρ and other sequences; 5. With 5-year follow-up data.

Exclusion Criteria:

* 1. Patients who are unable to undergo MRI scanning due to claustrophobia, abnormal renal function, etc.; 2. Patients who have undergone liver surgery in the past; 3. Patients with major diseases such as heart failure and tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease who may develop liver cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
HCC incidence rate | 5 years
  Rate of HCC among enrolled patients

CONTACTS AND LOCATIONS:
Overall Officials: Yaqin Zhang, MD, Ph.D, Study Chair — Fifth Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Yaqin, Zhang, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No